CLINICAL TRIAL: NCT05517551
Title: The Effect of Low-flow and Normal-flow Desflurane Anesthesia on Respiratory Parameters in Robotic-assisted Radical Prostatectomy
Brief Title: Comparison of Low and Normal Flow Anesthesia in Robotic Assisted Radical Prostatectomy
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Principal Investigator, Betül Güven, Principle Investigator, Ankara City Hospital Bilkent
Other Study IDs: E1-22-2755
Record Dates: First submitted 2022-08-23; First posted 2022-08-26 (Actual); Last update posted 2022-08-26 (Actual); Status verified 2022-08

CONDITIONS: Low Flow Anesthesia; Normal Flow Anesthesia; Robotic Surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- normal flow anesthesia: A fresh gas flow of 3 L/min will be applied continuously
  Interventions: Procedure: robotic assisted radical prostatectomy
- low flow anesthesia: A fresh gas flow of 3 L/min will be applied for the first 20 minutes after intubation , and then it will be reduced to 1 L/min.
  Interventions: Procedure: robotic assisted radical prostatectomy

INTERVENTIONS:
Procedure: robotic assisted radical prostatectomy — Patients who will undergo robotic-assisted laparoscopic prostatectomy surgery

SUMMARY:
Robot-assisted laparoscopic radical prostatectomy has gained increasing popularity compared to open radical prostatectomy with its advantages such as low blood loss, reduced blood transfusion rate, low complication rate, and shortened hospital stay. Since robot-assisted laparoscopic radical prostatectomy should be performed in the limited retroperitoneal area, insufflation of the abdomen with carbon dioxide (CO2) (pneumoperitoneum) and steep Trendelenburg position are required to provide better surgical vision.

Low-flow anesthesia warms and moistens the inhaled gases, creating a more physiological breathing atmosphere during anesthesia. In addition, it provides cost advantage by reducing inhalation agent consumption and reduces atmospheric pollution. Studies show that long-term minimal flow anesthesia is safe and advantageous for non-laparoscopic surgery.

The aim of this study is to compare low-flow (1L/min) with normal flow (3lt/min) desflurane anesthesia in terms of hemodynamic and respiratory parameters, inhalation agent consumption and soda lime consumption for robotic assisted laparoscopic radical prostatectomy surgery.

The secondary aim of the study is to compare the effects of low-flow and normal-flow anesthesia in the steep trendelenburg position (45°) used for robotically assisted laparoscopic radical prostatectomy.

ELIGIBILITY:
Inclusion Criteria:

- ASA I-II risk group

Exclusion Criteria:

* ASA III, IV, V,
* concomitant serious cardiac, respiratory, hepatic, renal disturbance,
* mental status disorder and hearing problem,
* anxiety and depression and/or other psychiatric disorders,
* patient's refusal

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients who will undergo robotic-assisted laparoscopic prostatectomy surgery
Sampling Method: Probability Sample
Enrollment: 68 (Estimated)
Dates: Start 2022-08 (Estimated); Primary Completion 2022-09 (Estimated); Study Completion 2023-03 (Estimated)

PRIMARY OUTCOMES:
inspiratory O₂ concentration | from beginning of anesthesia induction to the end of anesthesia (during periopertaive period)
  inspiratory O₂ concentration is measured from anesthesia machine monitor
partial oxygen pressure | from beginning of anesthesia induction to the end of anesthesia (during periopertaive period)
  PO2 from blood gas analysis

SECONDARY OUTCOMES:
desflurane consumption | perioperative
  desflurane consumption at the end of anesthesia is measured from anesthesia machine monitor
changes in liver and kidney function tests from the preoperative values to 48 hours postoperative | during operation and 48 hours postoperative
  to determine the changes in serum aspartate aminotransferase (AST), alanine aminotransferase (ALT), blood urea nitrogen (BUN), and creatinine from the preoperative values to 48 hours postoperative

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara City Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided